CLINICAL TRIAL: NCT03377725
Title: Decitabine and Arsenic Trioxide(ATO) in the Treatment of Myelodysplasic Syndrome
Brief Title: Decitabine and Arsenic Trioxide for Myelodysplastic Syndrome(MDS)
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: No patient was involved.
Sponsor: Li Junmin (Other)
Responsible Party: Sponsor-Investigator, Li Junmin, director of the hematology department, Ruijin Hospital
Organization: Ruijin Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RuijinH mutant p53 MDS
Record Dates: First submitted 2017-12-13; First posted 2017-12-19 (Actual); Last update posted 2023-08-16 (Actual); Status verified 2018-01

CONDITIONS: Myelodysplastic Syndromes; P53 Mutation
Keywords: Myelodysplastic Syndromes; Decitabine; Arsenic Trioxide; P53 Mutations
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — Decitabine; Arsenic Trioxide; Arsenic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): MDS patients of the experimental group will be treated with decitabine and arsenic trioxide.
  Interventions: Drug: Decitabine; Drug: Arsenic Trioxide
- Controlled group (Active Comparator): MDS patients of the controlled group will be treated with decitabine alone.
  Interventions: Drug: Decitabine

INTERVENTIONS:
Drug: Decitabine — 20mg/m^2,d1-5,ivgtt,28days as a duration
  Other Names: DNA demethylation agent; DNA damaging agent
Drug: Arsenic Trioxide — 0.16mg/kg,d1-5,ivgtt,28days as a duration
  Other Names: As2O3; Arsenic
  Arms: Experimental group

SUMMARY:
This is a prospective,controlled and multi-institution trial.The aim is to identify if using decitabine and Arsenic Trioxide(ATO) as the therapy of Myelodysplastic Syndrome(MDS) has better relapse free survival and complete response than using decitabine alone.

TP53 mutation is commonly associated with poor cancer patient prognosis yet no mutant p53 (mp53)-targeting regimen was clinically established. Particularly, p53 mutation is associated with extremely poor prognosis in myelodysplastic syndromes (MDS) and acute myeloid leukemia (AML) patients.

Decitabine (DAC) is a FDA approved drug for MDS treatment. In two independent clinical trials reported recently, DNA demethylating drug DAC treatment yielded a surprisingly high rate of complete remission (CR) in mp53-harboring AML/MDS patients (Welch, NEJM, 2016; Chang, BJH, 2017). Notably, all of the mp53-expressing patients in the two clinical studies relapsed quickly.

Arsenic trioxide (ATO) is a FDA approved drug for M3-AML treatment. Despite of the observed efficacy in treating non-APL patients, ATO is not yet approved for non-APL cancer treatment. ATO plays key role in regulating both wild-type p53 (wtp53) and mp53. Our published and unpublished data suggest ATO potentially hijacks nuclear iASPP-mediated STRaND pathway via exposing iASPP's RaDAR nuclear import code (Lu, Cancer Cell, 2013; Lu, Cell, 2014; Lu, Nat Rev Mol Cell Biol, 2016; Lu, unpublished). Our unpublished data also suggests a key role of ATO in regulating mp53 (Lu, The 17th International p53 Workshop, 2017). ATO is widely reported to be able to degrade and thus inhibit mp53's oncogenic function (Hamadeh, BBRC, 1999)(Liu, Blood, 2003). ATO suppressed cancer cell growth by targeting mp53 for degradation by Pirh2 degradation pathway (Yang, JBC, 2011; Yan, PLOS one, 2014);

Here we explore the potential of combination of DAC and ATO in improving the mp53-harboring AML/MDS patients' relapse free survival (RFS) and the ability to thoroughly eliminate mp53 subclone. Basic researches aiming to explore the mechanisms how mp53 cells responds to DAC and/or ATO treatment and how mp53 cells develop resistance to DAC and/or ATO will be coupled. We designate trials aiming for a better treatment regimen for mp53 patients as 'PANDA-Trials'.

DETAILED DESCRIPTION:
300 MDS patients will be recruited for trial. They will be randomly administrated with ATO + decitabine (n=200) or decitabine alone (n=100). The RSF, CR ratio, overall survival will be compared between the two arms. Importantly, TP53 status will be sequenced and its correlation with RSF, CR ratio, overall survival within the two arms will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* de novo MDS
* The Revised International Prognostic Scoring System(IPSS-R) is intermediate,poor or very poor
* 18-75years old(including 18-year-old and 75-year-old patients)
* ECOG<3,CCI≤1,ADL≥100
* bone marrow is active
* normal hepatic function and renal function
* normal cardiac function
* obtain informed consent

Exclusion Criteria:

* previously treated MDS patients
* abnormal hepatic function or renal function
* severe cardiac disease,including myocardial infarction,cardiac dysfunction
* ECG:QTc>0.44 sec in men,QTc>0.46 sec in women
* with other malignant tumor meanwhile
* active tuberculosis or HIV-positive patients
* woman who are pregnant or breastfeeding
* allergic to any drug in protocol or with contraindications
* hypomethylation agent(HMA) is contraindicated
* ECOG≥3,CCI>1,ADL<100
* cannot understand or obey the protocol
* with a history of allergies or intolerability
* with a history of decitabine therapy
* participate in other clinical trials meanwhile
* any situations that hinder trial existed

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-03-20 (Actual); Primary Completion 2018-03-31 (Actual); Study Completion 2018-03-31 (Actual)

PRIMARY OUTCOMES:
relapse free survival | up to 6-8 months after complete release
  since a patient first being determined as complete release until relapse

SECONDARY OUTCOMES:
complete release | 2-4 months since the first cycle of treatment
  the percent of patients with complete release in all patients enrolled
overall survival | primary estimated for 1year
  from first diagnosed to death whichever the cause is

CONTACTS AND LOCATIONS:
Overall Officials: Zhang Sujiang, Principal Investigator — Shanghai Ruijin Hospital North; Lu Min, Principal Investigator — Shanghai institute of Hematology
Locations (3):
- China (3):
  - Ruijin Hospital North, Shanghai
  - Ruijin Hospital, Shanghai
  - Shanghai Institute of Hematology, Shanghai

REFERENCES:
- [Background] Chang CK, Zhao YS, Xu F, Guo J, Zhang Z, He Q, Wu D, Wu LY, Su JY, Song LX, Xiao C, Li X. TP53 mutations predict decitabine-induced complete responses in patients with myelodysplastic syndromes. Br J Haematol. 2017 Feb;176(4):600-608. doi: 10.1111/bjh.14455. Epub 2016 Dec 16. PMID 27984642
- [Background] Welch JS, Petti AA, Miller CA, Fronick CC, O'Laughlin M, Fulton RS, Wilson RK, Baty JD, Duncavage EJ, Tandon B, Lee YS, Wartman LD, Uy GL, Ghobadi A, Tomasson MH, Pusic I, Romee R, Fehniger TA, Stockerl-Goldstein KE, Vij R, Oh ST, Abboud CN, Cashen AF, Schroeder MA, Jacoby MA, Heath SE, Luber K, Janke MR, Hantel A, Khan N, Sukhanova MJ, Knoebel RW, Stock W, Graubert TA, Walter MJ, Westervelt P, Link DC, DiPersio JF, Ley TJ. TP53 and Decitabine in Acute Myeloid Leukemia and Myelodysplastic Syndromes. N Engl J Med. 2016 Nov 24;375(21):2023-2036. doi: 10.1056/NEJMoa1605949. PMID 27959731
- [Background] Lu M, Breyssens H, Salter V, Zhong S, Hu Y, Baer C, Ratnayaka I, Sullivan A, Brown NR, Endicott J, Knapp S, Kessler BM, Middleton MR, Siebold C, Jones EY, Sviderskaya EV, Cebon J, John T, Caballero OL, Goding CR, Lu X. Restoring p53 function in human melanoma cells by inhibiting MDM2 and cyclin B1/CDK1-phosphorylated nuclear iASPP. Cancer Cell. 2013 May 13;23(5):618-33. doi: 10.1016/j.ccr.2013.03.013. Epub 2013 Apr 25. PMID 23623661
- [Background] Lu M, Muers MR, Lu X. Introducing STRaNDs: shuttling transcriptional regulators that are non-DNA binding. Nat Rev Mol Cell Biol. 2016 Aug;17(8):523-32. doi: 10.1038/nrm.2016.41. Epub 2016 May 25. PMID 27220640
- [Background] Lu M, Zak J, Chen S, Sanchez-Pulido L, Severson DT, Endicott J, Ponting CP, Schofield CJ, Lu X. A code for RanGDP binding in ankyrin repeats defines a nuclear import pathway. Cell. 2014 May 22;157(5):1130-45. doi: 10.1016/j.cell.2014.05.006. PMID 24855949
- [Background] Yan W, Jung YS, Zhang Y, Chen X. Arsenic trioxide reactivates proteasome-dependent degradation of mutant p53 protein in cancer cells in part via enhanced expression of Pirh2 E3 ligase. PLoS One. 2014 Aug 12;9(8):e103497. doi: 10.1371/journal.pone.0103497. eCollection 2014. PMID 25116336